CLINICAL TRIAL: NCT05152602
Title: Effect of Bilateral and Unilateral Erector Spinae Plane Block on Postoperative Pain in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Comparation of Bilateral and Unilateral Erector Spinae Plane Block
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-21-228
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain, Acute; Regional Anesthesia; Multimodal Analgesia
Keywords: ESP block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unilateral ESP block group: The group who underwent laparoscopic cholecystectomy and underwent unilateral ESP block for postoperative analgesia.
  Interventions: Procedure: Unilateral Erector spinae plane block
- Bilateral ESP block group: The group who underwent laparoscopic cholecystectomy and underwent bilateral ESP block for postoperative analgesia.
  Interventions: Procedure: Bilateral Erector spinae plane block
- Control group: The group that underwent laparoscopic cholecystectomy and underwent 1mg/kg tramadol and 50mg dexketoprofen for postoperative pain.

INTERVENTIONS:
Procedure: Bilateral Erector spinae plane block — Erector spinae plane (ESP) block is an interfascial plane block where a local anaesthetic is injected in a plane preferably below the erector spinae muscle. It is supposed to work at the origin of spinal nerves based on cadaveric and contrast study. It has emerged as an effective and safe analgesic regional technique. It will be done at T7-8 level
  Groups: Bilateral ESP block group
Procedure: Unilateral Erector spinae plane block — Erector spinae plane (ESP) block is an interfascial plane block where a local anaesthetic is injected in a plane preferably below the erector spinae muscle. It is supposed to work at the origin of spinal nerves based on cadaveric and contrast study. It has emerged as an effective and safe analgesic regional technique. It will be done at T7-8 level
  Groups: Unilateral ESP block group

SUMMARY:
Although laparoscopic cholecystectomy is a minimally invasive surgery with many advantages, it is one of the operations with high postoperative pain scores. Opioids are frequently used to prevent postoperative pain. Due to the side effects of opioids, the amount of use is tried to be reduced. Regional anesthesia techniques can be used to minimize opioid consumption. Erector spina plane block was first described in 2016 by Forero et al. in the treatment of thoracic neuropathic pain. Since then, ESP block has been used as an anesthetic and analgesic technique. It is applied by injecting local anesthetic into the fascial plane located between the erector spina muscle and the transverse process of the vertebra. Several high-level studies have shown that the ESP block can be used to reduce postoperative pain after gastrointestinal surgery. Several studies have evaluated the effect of ESP block for pain relief after laparoscopic cholecystectomy. ESP block has been applied unilaterally or bilaterally in various studies. However, in the current studies in the literature, the advantages or disadvantages of the bilateral application of the ESP block compared to the unilateral application have not been evaluated. In this study, the investigators aimed to evaluate postoperative pain by applying ESP block to patients who underwent laparoscopic cholecystectomy and to evaluate the advantages of unilateral or bilateral application of ESP block over each other.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent laparoscopic cholecystectomy surgery between December 2021 and January 2022 will participate in the study.

Exclusion Criteria:

* There is no exclusion criteria for the study.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients who had laparoscopic cholecystectomy between December 2021 and January 2022.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 0-24 hour
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Opioid consumption | 24 hour
  Total usage of opioid's dosage when the patients VAS scores over than the four

CONTACTS AND LOCATIONS:
Overall Officials: Ayça T. Dumanlı Özcan, Assoc. Prof., Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang J, Liu JC. Ultrasound-guided erector spinae plane block for postoperative analgesia: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 Apr 14;20(1):83. doi: 10.1186/s12871-020-00999-8. PMID 32290814
- [Result] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Sercan O, Karaveli A, Ozmen S, Uslu A. Comparison of the Effects of Pectoral Nerve Block and Local Infiltration Anesthesia on Postoperative Pain for Breast Reduction Surgery: A Prospective Observational Study. Eurasian J Med. 2021 Jun;53(2):102-107. doi: 10.5152/eurasianjmed.2021.20111. PMID 34177291